CLINICAL TRIAL: NCT04847570
Title: The Effect of Music on Patients in Critical Care (EMPIRE)
Brief Title: The Effect of Music on Patients in Critical Care
Acronym: EMPIRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Collaborators: CW+ Charity (Other); Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C&W21/009
Record Dates: First submitted 2021-03-25; First posted 2021-04-19 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Intensive Care
Keywords: Music; AICU; Inpatient

STUDY DESIGN:
Intervention Model Description: Non-clinical intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music listening experience (Experimental): It is a single-arm non-randomised study. The same inclusion and exclusion criteria applies to all the participants.
  Interventions: Other: Music session

INTERVENTIONS:
Other: Music session — Non-clinical intervention only, and no change to clinical care or treatment. Participants will have 10 minutes of undisturbed rest, followed by a supervised music-listening session of up to 40 minutes, ending with another 10-minute rest period.

SUMMARY:
The EMPIRE study will assess the effect of music listening on patients in critical care. 30 patients from the Adult Intensive Care Unit (AICU) at Chelsea and Westminster Hospital will be recruited to undergo a single 40-minute session of supervised music listening. Before and after the session, patients will be asked to describe their pain and anxiety on a rating of 1-10, and the patient's level of agitation/sedation will also be measured. In addition, physiological data such as heart rate, respiratory rate, blood pressure and level of sedation (bispectral index score) will be measured throughout the listening session. Finally, a 3-month follow-up interview will be conducted to assess the influence of the music on participants' experience of the Adult Intensive Care Unit.

DETAILED DESCRIPTION:
The EMPIRE study will assess the effect of music listening on patients in critical care. Treatment on an intensive care unit can be disorientating and frightening, with patients at risk of delirium and post-traumatic stress disorder. The COVID-19 pandemic has exacerbated some of the factors which might contribute to this, such as lack of visits from relatives and friends, increased difficulty communicating with staff, and an increased likelihood of being on mechanical ventilation and sedation. Music has shown the potential to be a low-cost non-pharmacological intervention which can improve patients' experience of acute care without adding significantly to the workload of staff.

Studies have suggested that music listening has the potential to reduce feelings of pain and anxiety in critical care patients, as well as improved autonomic physiological outcomes such as heart rate, respiratory rate and blood pressure.

The EMPIRE study will seek to explore the effects described above in greater detail. 30 patients from the Adult Intensive Care Unit (AICU) at Chelsea and Westminster Hospital will be recruited to undergo a single 40-minute session of supervised music listening, in which they will be encouraged to request their favourite music if they are able. Before and after the session, patients will be asked to describe their pain and anxiety on a rating of 1-10, and the patient's level of agitation/sedation will also be measured, so that changes in these can be evaluated. In addition, physiological data such as heart rate, respiratory rate, blood pressure and level of sedation (bispectral index score) will be measured throughout the listening session, and later analysed for significant changes in relation to the music that was being played. Finally, a 3-month follow-up interview will be conducted to assess the influence of the music on participants' experience of the Adult Intensive Care Unit.

ELIGIBILITY:
Inclusion Criteria:

* Nominated for participation by the clinical team of the Chelsea and Westminster Hospital AICU
* Level 1-3 critical care inpatient at Chelsea and Westminster Hospital AICU
* Age 18 or above
* English speaking
* RASS score >-2
* No significant hearing loss (able to hear music being played)
* Consent obtained from patient or advice sought from consultee (personal or nominated (professional))

Exclusion Criteria:

* Under 18 years of age
* Non-English speaking
* RASS score <-2
* Significant hearing loss (not able to hear music being played)
* Unable to obtain consent from patient or receive advice from consultee (personal or nominated)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-10-04 (Estimated); Study Completion 2021-10-04 (Estimated)

PRIMARY OUTCOMES:
Investigate the effect of music on state anxiety | 6 months
  Verbal anxiety rating, 0-10, pre/post.
Investigate the effect of music on pain | 6 months
  Either ONRS 0-10, or C-POT 0-8, pre/post
Investigate the effect of music on agitation | 6 months
  RASS, -5 to +4, pre-/post
Investigate the effect of music on HR | 6 months
  Measured in beats per minute
Investigate the effect of music on RR | 6 months
  Measured in breaths per minute
Investigate the effect of music on DBP and SBP | 6 months
  Measured in mm Hg
Investigate the effect of music on BIS | 6 months
  Measured using the Bispectral index (BIS)
Investigate the longitudinal effects of music on ICU experience | 3 months
  Follow up interview 3 months later

SECONDARY OUTCOMES:
Correlation analysis of continuous HR, RR, BP and BIS data with the following musical analysis data (drawn from the Spotify API): | 6 months
  * Acousticness (0-1)
  * Danceability (0-1)
  * Duration (continuous)
  * Energy (0-1)
  * Instrumentalness (0-1)
  * Key (0-11)
  * Liveness (0-1)
  * Loudness (db, c.-60 to 0)
  * Mode (0-1)
  * Speechiness (0-1)
  * Tempo (continuous)
  * Time Signature (continuous)
  * Valence (0-1)

CONTACTS AND LOCATIONS:
Locations (1):
- Chelsea and Westminster Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ames N, Shuford R, Yang L, Moriyama B, Frey M, Wilson F, Sundaramurthi T, Gori D, Mannes A, Ranucci A, Koziol D, Wallen GR. Music Listening Among Postoperative Patients in the Intensive Care Unit: A Randomized Controlled Trial with Mixed-Methods Analysis. Integr Med Insights. 2017 Jul 20;12:1178633717716455. doi: 10.1177/1178633717716455. eCollection 2017. PMID 28904523
- [Background] Benotsch EG, Lutgendorf SK, Watson D, Fick LJ, Lang EV. Rapid anxiety assessment in medical patients: evidence for the validity of verbal anxiety ratings. Ann Behav Med. 2000 Summer;22(3):199-203. doi: 10.1007/BF02895114. PMID 11126464
- [Background] Bradt J, Dileo C. Music interventions for mechanically ventilated patients. Cochrane Database Syst Rev. 2014;2014(12):CD006902. doi: 10.1002/14651858.CD006902.pub3. Epub 2014 Dec 9. PMID 25490233
- [Background] Cardoso, L. et al. (2017) 'Music therapy as an autonomous intervention of nurses for pain control in icu: integrative review', Millenium - Journal of Education, Technologies, and Health, 2(04), pp. 89-100. doi: 10.29352/mill0204.08.00148.
- [Background] Chanques G, Viel E, Constantin JM, Jung B, de Lattre S, Carr J, Cisse M, Lefrant JY, Jaber S. The measurement of pain in intensive care unit: comparison of 5 self-report intensity scales. Pain. 2010 Dec;151(3):711-721. doi: 10.1016/j.pain.2010.08.039. Epub 2010 Sep 16. PMID 20843604
- [Background] Chlan LL, Engeland WC, Anthony A, Guttormson J. Influence of music on the stress response in patients receiving mechanical ventilatory support: a pilot study. Am J Crit Care. 2007 Mar;16(2):141-5. PMID 17322014
- [Background] Davydow DS, Gifford JM, Desai SV, Needham DM, Bienvenu OJ. Posttraumatic stress disorder in general intensive care unit survivors: a systematic review. Gen Hosp Psychiatry. 2008 Sep-Oct;30(5):421-34. doi: 10.1016/j.genhosppsych.2008.05.006. Epub 2008 Jul 30. PMID 18774425
- [Background] Gelinas C, Fillion L, Puntillo KA, Viens C, Fortier M. Validation of the critical-care pain observation tool in adult patients. Am J Crit Care. 2006 Jul;15(4):420-7. PMID 16823021
- [Background] Han L, Li JP, Sit JW, Chung L, Jiao ZY, Ma WG. Effects of music intervention on physiological stress response and anxiety level of mechanically ventilated patients in China: a randomised controlled trial. J Clin Nurs. 2010 Apr;19(7-8):978-87. doi: 10.1111/j.1365-2702.2009.02845.x. PMID 20492042
- [Background] Jafari H, Emami Zeydi A, Khani S, Esmaeili R, Soleimani A. The effects of listening to preferred music on pain intensity after open heart surgery. Iran J Nurs Midwifery Res. 2012 Jan;17(1):1-6. PMID 23493927
- [Background] Kyavar, M. et al. (2016) 'Effect of preferred music listening on pain reduction in mechanically ventilated patients after coronary artery bypass graft surgery', Research in Cardiovascular Medicine, 5(4), p. 8. doi: 10.5812/cardiovascmed.33769.
- [Background] Lee CH, Lee CY, Hsu MY, Lai CL, Sung YH, Lin CY, Lin LY. Effects of Music Intervention on State Anxiety and Physiological Indices in Patients Undergoing Mechanical Ventilation in the Intensive Care Unit. Biol Res Nurs. 2017 Mar;19(2):137-144. doi: 10.1177/1099800416669601. Epub 2016 Sep 21. PMID 27655993
- [Background] Lee OK, Chung YF, Chan MF, Chan WM. Music and its effect on the physiological responses and anxiety levels of patients receiving mechanical ventilation: a pilot study. J Clin Nurs. 2005 May;14(5):609-20. doi: 10.1111/j.1365-2702.2004.01103.x. PMID 15840076
- [Background] Nilsson U. The anxiety- and pain-reducing effects of music interventions: a systematic review. AORN J. 2008 Apr;87(4):780-807. doi: 10.1016/j.aorn.2007.09.013. PMID 18395022
- [Background] Richard-Lalonde M, Gelinas C, Boitor M, Gosselin E, Feeley N, Cossette S, Chlan LL. The Effect of Music on Pain in the Adult Intensive Care Unit: A Systematic Review of Randomized Controlled Trials. J Pain Symptom Manage. 2020 Jun;59(6):1304-1319.e6. doi: 10.1016/j.jpainsymman.2019.12.359. Epub 2019 Dec 24. PMID 31881291
- [Background] Samuelson KA. Unpleasant and pleasant memories of intensive care in adult mechanically ventilated patients--findings from 250 interviews. Intensive Crit Care Nurs. 2011 Apr;27(2):76-84. doi: 10.1016/j.iccn.2011.01.003. Epub 2011 Mar 2. PMID 21371888
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Background] Stratton, V. N. and Zalanowski, A. H. (1984) 'The relationship between music, degree of liking, and self-reported relaxation', Journal of Music Therapy, 21(4), pp. 184-192. doi: 10.1093/jmt/21.4.184.